CLINICAL TRIAL: NCT05546463
Title: The Effects of Playing Digital Games on Children's Pain, Fear and Anxiety Levels During Suturing: A Randomized Controlled Study
Brief Title: The Effects of Playing Digital Games on Children's Pain, Fear and Anxiety Levels During Suturing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Tülay YAVAN, Prof, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IzmirUEcon
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pain, Procedural; Fear of Needles; Anxiety State
MeSH Terms: conditions — Pain, Procedural; Iatrophobia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): During the suture procedure, the children in the intervention group played digital games.
  Children began playing digital games about one minute before the local anesthesia procedure, continued to play digital games throughout the suturing procedure.
  Interventions: Behavioral: Digital games
- Control group (Experimental): During the suture procedure, the children in the control group did not play digital games.
  Interventions: Behavioral: Digital games

INTERVENTIONS:
Behavioral: Digital games — A digital game was played via iPad Air 2 32GB 9.7-inch wi-fi model tablet. The researcher created a folder with a range of selected games to appeal to different preferences. Children could choose from the following games: Word Travel, Talking Tom Candy Run, 384 Puzzles for Kids, Masha and The Bear, Subway Surfers, Head Ball 2 and Dream League Soccer".

SUMMARY:
The aim was to determine the effects of digital game play on children's pain, fear and anxiety levels during suturing.

Data was obtained from 84 children between the ages of 8-17 at the Pediatric Emergency Department between 16 January and 19 March 2020, using the Socio-Demographic and Clinical Characteristics Form, the Wong-Baker Faces Pain Rating Scale (WBFPS), the Visual Analogue Scale (VAS), the Fear of Medical Procedure Scale (FMPS), and the State-Trait Anxiety Inventory for Children (STAI-CH). While the study group (n=42) played digital games during the suturing procedure, the control group (n=42) did not play digital games.

DETAILED DESCRIPTION:
This study has the potential to contribute to the literature on the effects of playing digital games on the pain, fear, and anxiety levels that children experience during suturing.

Materials and Methods

Design, setting, and sample size:

The data of the randomized controlled study were collected in the Pediatric Emergency Department (PED) of the Training and Research Hospital between 16 January and 19 March 2020. The population of the study are children between the ages of 8 and 17 who were sutured in the PED. Random sampling method was used for participant selection. The size of the sample was determined by the power analysis of the GPower 3.1.9.4 program as 84 children with 0.05 error, 0.95 confidence interval, and 0.5 effect size.

Participants and randomization:

The inclusion criteria were that children were between the ages of 8-17 and had no psychological diagnoses, had no problems in vision, hearing, or speech, spoke and understood Turkish, that the number of sutures was 3 or more (generally, local anesthesia is not applied to 1-2 sutures), that the suture procedure was performed under local anesthesia, and that they assented to participate in the study. Exclusion criteria were refusing to play digital games or stop playing before the process ends, having a physical problem that prevents playing digital games, being too agitated to communicate with the child. Children were divided into two groups (intervention group: n=42 and control group: n=42), using the block of four randomization methods among those who met the inclusion criteria, according to their order of admission to the PED. The children in the intervention and control groups did not know which group they were in and did not encounter each other. First researcher is staff member within the PED, and performed the randomization.

Ethical Approach:

Permission was obtained from Ethics Committee of University (Issue No: excluded double-blind review) and the institution where the research would be conducted (Date:15/01/2020). Original signed consent was obtained from all parents who assented to participate in the study through the Information and Informed Consent Form. Verbal consent was obtained from the children assented. A health professional acting as a witness signed a form to this effect.

Data Collection Tools:

Research data were collected using "Socio-Demographic and Clinical Characteristics Form", "Wong-Baker Faces Pain Rating Scale", "Visual Analogue Scale", "State-Trait Anxiety Inventory for Children", and "Fear for Medical Procedures Scale". First researcher informed the children and their parents about the tools, and collect the data. The average data collection time was 30 minutes. Data were obtained using face-to-face interviews and observation from children.

Socio-Demographic and Clinical Characteristics Form:

This form consists of a total of 23 questions eliciting information, including on age, gender, previous digital game playing status, number of suturing, and duration of suturing, created by the researchers in accordance with the literature.

Wong-Baker Faces Pain Rating Scale (WBFPS):

The Faces Pain Rating Scale, developed by Wong and Baker, is a hand-drawn scale that includes six facial expressions ranging from smiling to crying, and is recommended for use for children aged 3 years and older. Scoring is defined as 0 = no hurt, 2 = hurts little bit, 4 = hurts little more, 6 = hurts even more, 8 = hurts whole lot, 10 = hurts worst.

Visual Analogue Scale (VAS):

This is a 100 mm long horizontal line with the words "no pain" and "severe pain" at either end. It is suitable for school-age children. The child is asked to mark the point showing the intensity of pain felt at that moment.

Fear of Medical Procedures Scale:

Fear of Medical Procedures Scale (FMPS) was developed by Bloom et al. in 1985 to assess children's fears associated with medical procedures and practices. The scale consists of 29 questions evaluating the fear of medical procedures. The scale consists of 4 sub-dimensions, including operational, personal, environmental, and interpersonal items. In the three-point Likert-type scale, for each question, children are asked to choose one of the expressions "no fear" (1 point), "moderate fear" (2 points), "high fear" (3 points). Scores range between 29 and 87. The validity and reliability study in Türkiye was conducted among children aged 7-14 by Alak in 1993, and the reliability coefficient was found to be .93. In our study, the Cronbach Alpha value of the scale was found to be .93.

State-Trait Anxiety Inventory for Children:

State-Trait Anxiety Inventory for Children (STAI-CH) was developed by Spielberger in 1973 to measure the anxiety caused to children in particular situations perceived as a threat. In the trait anxiety scale, the children are asked to evaluate how they "generally" feel, and in the state anxiety scale, how they feel in the situation they are in "at that moment", and indicate one of three options. Possible scores range between 20 and 60. A higher score indicates greater anxiety. The validity and reliability study in Türkiye was conducted by Özusta in 1995 for children aged 9-12. In STAI-CH, the Cronbach Alpha coefficient of the state anxiety scale was found .82, and the Cronbach Alpha coefficient of the trait anxiety scale was .81. In our study, the Cronbach Alpha coefficient of the state anxiety scale was found .91, and the Cronbach Alpha coefficient of the trait anxiety scale was .78.

Procedure:

A digital game was played via iPad Air 2 32GB 9.7-inch wi-fi model tablet. The researcher created a folder with a range of selected games to appeal to different preferences. Children could choose from the following games: Word Travel, Talking Tom Candy Run, 384 Puzzles for Kids, Masha and The Bear, Subway Surfers, Head Ball 2 and Dream League Soccer".

During the suture procedure, the children in the intervention group played digital games, while the children in the control group did not. The routine practices of the clinic were carried out in both groups.

In the pre-procedure, the researcher completed the Socio-Demographic and Clinical Characteristics Form, with an explanation about WBFPS, VAS, FMPS, and STAI-CH. Families were allowed to stay with their children. Children in the intervention group began playing digital games about one minute before the local anesthesia procedure (Figure 1).

The children in the intervention group continued to play digital games throughout the suturing procedure. Children in all groups were asked to mark the pain they experienced during the procedure on the WBFPS and VAS. Parents were encouraged to stand next to the child during the process.

In post-procedure, children in all groups were asked to mark the pain experienced after suturing on the WBFPS and VAS. All children were asked to respond to the FMPS and STAI-CH (only state inventory) scales to measure the fear and anxiety experienced.

Statistical Analysis:

Licensed SPSS (Statistical Package for the Social Science) for Windows 25.0.0 package program was used for data analysis. The suitability of the data to the normal distribution was examined with the Kolmogorov-Smirnov test. Continuous variables are expressed as mean ± standard deviation. According to the results of the normality test, either the t-test or Mann-Whitney U test was used in independent groups for comparisons between groups. Intergroup comparisons of categorical variables, as for that, were performed using Pearson Chi-square test or Fisher Exact test. In group comparisons, t-test, Wilcoxon test, and multiple analysis of variance were used in repeated measurements in dependent groups. Tukey's test was used for Post-Hoc analysis with Bonferroni correction to determine which group caused the difference. The results were evaluated at a 95% confidence interval and p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Having no psychological diagnoses.
* Having no problems in vision, hearing, or speech.
* Speaking and understanding Turkish.
* That the number of sutures is 3 or more.
* That the suture procedure is performing under local anesthesia.
* That they assent to participate in the study.

Exclusion Criteria:

* Refusing to play digital games or stop playing before the process ends.
* Having a physical problem that prevents playing digital games.
* Being too agitated to communicate with the child.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Socio-Demographic and Clinical Characteristics | 2 months
  Socio-Demographic and Clinical Characteristics Form:
  This form consists of a total of 23 questions eliciting information, including on age, gender, previous digital game playing status, number of suturing, and duration of suturing, created by the researchers in accordance with the literature.
Pain score | 2 months
  Pain score was determined using "Wong-Baker Faces Pain Rating Scale" and "Visual Analogue Scale".
  Wong-Baker Faces Pain Rating Scale:
  The Faces Pain Rating Scale, developed by Wong and Baker, is a hand-drawn scale that includes six facial expressions ranging from smiling to crying, and is recommended for use for children aged 3 years and older. Scoring is defined as 0 = no hurt, 2 = hurts little bit, 4 = hurts little more, 6 = hurts even more, 8 = hurts whole lot, 10 = hurts worst.
  Visual Analogue Scale:
  This is a 100 mm long horizontal line with the words "no pain" and "severe pain" at either end. It is suitable for school-age children. The child is asked to mark the point showing the intensity of pain felt at that moment.
Anxiety score | 2 months
  Anxiety score was determined using "State-Trait Anxiety Inventory for Children"
  State-Trait Anxiety Inventory for Children:
  State-Trait Anxiety Inventory for Children was developed by Spielberger in 1973 to measure the anxiety caused to children in particular situations perceived as a threat. In the trait anxiety scale, the children are asked to evaluate how they "generally" feel, and in the state anxiety scale, how they feel in the situation they are in "at that moment", and indicate one of three options. Possible scores range between 20 and 60. A higher score indicates greater anxiety. The validity and reliability study in Türkiye was conducted by Özusta in 1995 for children aged 9-12. In State-Trait Anxiety Inventory for Children, the Cronbach Alpha coefficient of the state anxiety scale was found .82, and the Cronbach Alpha coefficient of the trait anxiety scale was .81.
Fear score | 2 months
  Fear score was determined using "Fear for Medical Procedures Scale".
  Fear of Medical Procedures Scale:
  Fear of Medical Procedures Scale was developed by Bloom et al. in 1985 to assess children's fears associated with medical procedures and practices. The scale consists of 29 questions evaluating the fear of medical procedures. The scale consists of 4 sub-dimensions, including operational, personal, environmental, and interpersonal items. In the three-point Likert-type scale, for each question, children are asked to choose one of the expressions "no fear" (1 point), "moderate fear" (2 points), "high fear" (3 points). Scores range between 29 and 87. The validity and reliability study in Türkiye was conducted among children aged 7-14 by Alak in 1993, and the reliability coefficient was found to be .93.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Ogce, Prof, Study Director — Izmir University of Economics
Locations (1):
- Health Sciences University Izmir Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)